CLINICAL TRIAL: NCT03845309
Title: The Effect of Using Nutrition Education as an Intervention Measure on Elevating the Nutritional Status, Quality of Life, and Self-Care Behavior of Patients With Chronic Heart Failure
Brief Title: Nutritional Interventions in Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201810039RINA
Record Dates: First submitted 2019-01-08; First posted 2019-02-19 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2020-12

CONDITIONS: Chronic Heart Failure; Nutrition
Keywords: Heart failure; Nutritional intervention; Quality of Life; Self-Care Behavior
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional intervention for CHF (Experimental)
  Interventions: Behavioral: Self-Care Behavior

INTERVENTIONS:
Behavioral: Self-Care Behavior — Limitations on liquid and sodium intake will be established in accordance with the NYHA functional classification, and patients will be provided with dietary assessments and nutrition advice according to personal characteristics such as age, physical activity level, and comorbidities. Additionally, suggestions on lifestyle changes were provided by referring to the advice for patients with heart failure from the American Heart Association.

SUMMARY:
This study recruited patients diagnosed with heart failure by cardiologists and cardiac outpatients whose cardiac functions were graded from 1 to 4 according to the New York Heart Association as the study participants. The participants were provided active nutrition intervention including diet optimization,specific recommendations and nutritional supplement prescriptions in cases in which nutritional goals were not reached.In addition, this study offered advice by referencing lifestyle change advice provided by the American Heart Association for patients with heart failure.

The Mini Nutritional Assessment Short-Form was used to assess malnutrition indicator values. The participant water, nutrient (i.e., carbohydrates, protein, and fat), and calorie intake data were collected using their recollection of their dietary intake and food intake frequency over a 24-hour dietary recall. The amount of fluid and sodium administered was provided according to the cardiac function grades indicated by the New York Heart Association.In addition, dietary assessments and nutritional advice were offered on the basis of the patients' conditions (i.e., age, activity, and comorbidity).

Finally, instrumental activities of daily living, EQ-5D (an instrument for measuring quality of life), grip performance, and 6-minute walk test data were utilized to analyze the changes in the participants before and after intervention, identifying the correlation between using nutrition education as an intervention measure and improvement in the participants' nutritional status, quality of life, and self-care behavior.

DETAILED DESCRIPTION:
Malnutrition may be caused by decreased nutrient intake or absorption, inflammation, or other disease-related mechanisms. Malnutrition resulting from disease or injury may be caused by decreased food intake or varying degrees of acute or chronic inflammation, which alters body composit ion and prompts a decline in biological functions. The effects of decreased food intake induced by an inflammatory reaction are related to the malnourishment resulted from anorexia, changes in metabolism, increased resting energy expenditure, and increased muscle catabolism. Changes in body composition are characterized by a decrease in any muscle mass marker (excluding fat mass, muscle mass index, or body cell mass). Therefore, malnutrition is associated with clinical results of clinical malfunction.

The primary objectives of heart failure treatment include preventing the need for hospitalization, increasing the survival rate, and improving health status. Patient symptoms, bodily functions, and health status are also referred to as health-related quality of life (HRQoL). The EuroQol-5D (EQ-5D) is used to assess the quality of life of patients undergoing cardiac rehabilitation. This assessment uses 5 aspects, namely mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, to assess patient health status.

Cardiopulmonary exercise testing (CPET) is the gold standard method for evaluating the motor ability of patients with chronic heart failure (CHF), yet is not extensively used. A more commonly used and simpler method is the 6-minute walk test, which measures the distance traveled by walking for 6 minutes. Changes in this value correlate to quality of life. This test is used to investigate the ability to perform daily activities and intensity of exercise in patients with mild to moderate CHF.

Muscle strength is a key indicator for assessing patients with sarcopenia because decreased muscle strength is considered a crucial element in diagnosing muscle reduction. For circumstances in which muscle mass is difficult to assess, muscle strength, such as handgrip strength, can serve as a standard assessment of muscle functions.

Exercise training is considered a valid method for stabilizing patients with heart failure. One study reported that the self-management intervention of a patient with heart failure notably decreased the occurrence of hospitalization and hospital readmission related to heart failure as well as all-cause mortality.

The present study determines the effectiveness of nutrition intervention in routine medical treatment for improving the nutrition and quality of care among patients with heart failure.

This study does not involve drugs, medical technology, or medical equipment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with CHF by a cardiologist. Clinical patients with the functional classification of NYHA FcI-NYHA FcⅣ according to the New York Heart Association (NYHA).
2. Adults aged 20 years or older who are conscious, have normal cognitive function, can walk without assistance, and do not require breathing aids. Additionally, participants must be able to answer questionnaires in Mandarin Chinese or Taiwanese, either orally or in writing.
3. Patients who have agreed to participate in the study by completing a consent form.

Exclusion Criteria:

1. Patients with an expected survival period of less than 6 months because of a disease not related to CHF
2. Long-term bed-bound patients
3. Patients with no potential for rehabilitation because of decline in functions of neural or musculoskeletal systems
4. Patients with severe disorders of consciousness or cognitive disorders or those with mental illness
5. Patients who require breathing aids for an extended period of time
6. Patients with end-stage severe CHF who have been diagnosed by doctors as unable to recover within a short period
7. Patients who are scheduled to undergo coronary artery bypass surgery or a heart valve surgery within 1 month
8. Patients who are on hemodialysis or are awaiting a kidney transplant
9. Patients with severe pulmonary diseases who require long-term home oxygen therapy
10. Patients who themselves decline to participate or who have a family member who objects to their participation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2020-12-13 (Actual)

PRIMARY OUTCOMES:
Mini Nutritional Assessment Short-Form | Change from Baseline Mini Nutritional Assessment Short-Form on months 0, 3 at 6 months(Do higher values represent a better outcome).
  Assess malnutrition indicator values. Nutrition status evaluated by the MNA correlates with energy and nutrient intakes as well as anthropometrics, hematologic, and biological nutrition parameters.
  MNA has 4 sections: anthropometrics (BMI, weight loss, arm and calf circumference), general assessment (lifestyle, medication, mobility, presence of depression or dementia), dietary assessment (number of meals, food and fluid intake, autonomy of feeding), and subjective assessment (self-perception of health and nutrition).
  The maximum score for the MNA-SF is 14, with scores ≥12 indicating satisfactory nutrition status and ≤11 indicating a risk of malnutrition.
Instrumental Activities of Daily Living | Change from Baseline Instrumental Activities of Daily Living on months 0, 3 at 6 months.
  Instrumental Activities of Daily Living Heath-related quality of life. IADL Scale was developed to assess more complex activities (termed "instrumental activities of daily living") necessary for functioning in community settings (e.g., shopping, cooking, managing finances). The capacity to handle these complex functions normally is lost before basic "activities of daily living" (e.g., eating, bathing, toileting) which are measured by ADL scales. Therefore, assessing IADLS may identify incipient decline in older adults or other individuals who are otherwise capable and healthy.
  It contains 8 items that are rated with a summary score from 0 (low functioning) to 8 (high functioning).
  This scale can be administered through an interview or by a written questionnaire.
EuroQol-5D | Change from Baseline EuroQol-5D on months 0, 3 at 6 months(Do higher values represent a better outcome).
  Assess the quality of life of patients undergoing cardiac rehabilitation. the generic EuroQol fivedimensional questionnaire (EQ-5D) instrument are commonly referred to as value sets; an important distinction lies in whether the valuations are elicited from individuals with experience of the health state (experience-based values) or from individuals from the general population to whom the health states are described (hypothetical values).
  * 100 means the best health you can imagine.
  * 0 means the worst health you can imagine.
Handgrip strength | Change from Baseline Handgrip strength on months 0, 3 at 6 months.
  Assessment of muscle functions. Measured by dynamometer, before and after intervention. We will compare the statistical properties of between baseline and after 0, 3 at 6 months intervention.
6-Minute walk test | Change from Baseline 6-Minute walk test on months 0, 3 at 6 months(Do higher values represent a better outcome).
  Changes in this value correlate to quality of life

SECONDARY OUTCOMES:
Energy intake | Change from Baseline Energy intake on months 0, 3 at 6 months.
  Energy intake (Kcal/day)will be assessed by dietary survey on 24-hour recall.
Carbohydrate intake | Change from Baseline Carbohydrate intake on months 0, 3 at 6 months.
  Carbohydrate intake (g / day) will be assessed by dietary survey on 24-hour recall.
Protein intake | Change from Baseline Protein intake on months 0, 3 at 6 months.
  Protein intake (g / day) will be assessed by dietary survey on 24-hour recall.
Fat intake | Change from Baseline Fat intake on months 0, 3 at 6 months.
  Fat intake (g / day) will be assessed by dietary survey on 24-hour recall.
Sodium intake | Change from Baseline Sodium intake on months 0, 3 at 6 months.
  Sodium intake (gm / day) will be evaluated by dietary survey on 24-hour recall.
Water intake | Change from Baseline Water intake on months 0, 3 at 6 months.
  Water intake (ml / day) will be evaluated by dietary survey on 24-hour recall.

CONTACTS AND LOCATIONS:
Overall Officials: Jien-Jiun Chen, MD, Principal Investigator — National Taiwan University Hospital; Feng-Ching Liao, BS, Principal Investigator — National Taiwan University Hospital; Sheng Nan Chang, PhD, Principal Investigator — National Taiwan University Hospital; Shao-Chi Yang, MD, Principal Investigator — National Taiwan University Hospital; Chih-Neng Hsu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Internal Medicine, National Taiwan Univeristy Hospital Yun-Lin branch, Douliu, Yunlin County, Taiwan

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data for all primary and secondary outcome meaurses will be made available

REFERENCES:
- [Background] Abshire M, Xu J, Baptiste D, Almansa JR, Xu J, Cummings A, Andrews MJ, Dennison Himmelfarb C. Nutritional Interventions in Heart Failure: A Systematic Review of the Literature. J Card Fail. 2015 Dec;21(12):989-99. doi: 10.1016/j.cardfail.2015.10.004. Epub 2015 Oct 23. PMID 26525961
- [Background] Jensen GL, Mirtallo J, Compher C, Dhaliwal R, Forbes A, Grijalba RF, Hardy G, Kondrup J, Labadarios D, Nyulasi I, Castillo Pineda JC, Waitzberg D; International Consensus Guideline Committee. Adult starvation and disease-related malnutrition: a proposal for etiology-based diagnosis in the clinical practice setting from the International Consensus Guideline Committee. JPEN J Parenter Enteral Nutr. 2010 Mar-Apr;34(2):156-9. doi: 10.1177/0148607110361910. PMID 20375423
- [Background] Anthony PS. Nutrition screening tools for hospitalized patients. Nutr Clin Pract. 2008 Aug-Sep;23(4):373-82. doi: 10.1177/0884533608321130. PMID 18682588
- [Background] Cederholm T, Barazzoni R, Austin P, Ballmer P, Biolo G, Bischoff SC, Compher C, Correia I, Higashiguchi T, Holst M, Jensen GL, Malone A, Muscaritoli M, Nyulasi I, Pirlich M, Rothenberg E, Schindler K, Schneider SM, de van der Schueren MA, Sieber C, Valentini L, Yu JC, Van Gossum A, Singer P. ESPEN guidelines on definitions and terminology of clinical nutrition. Clin Nutr. 2017 Feb;36(1):49-64. doi: 10.1016/j.clnu.2016.09.004. Epub 2016 Sep 14. PMID 27642056
- [Background] Soeters PB, Reijven PL, van Bokhorst-de van der Schueren MA, Schols JM, Halfens RJ, Meijers JM, van Gemert WG. A rational approach to nutritional assessment. Clin Nutr. 2008 Oct;27(5):706-16. doi: 10.1016/j.clnu.2008.07.009. Epub 2008 Sep 9. PMID 18783855
- [Background] Cederholm T, Jensen GL, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, Baptista G, Barazzoni R, Blaauw R, Coats A, Crivelli A, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren MAE, Siltharm S, Singer P, Tappenden K, Velasco N, Waitzberg D, Yamwong P, Yu J, Van Gossum A, Compher C; GLIM Core Leadership Committee; GLIM Working Group. GLIM criteria for the diagnosis of malnutrition - A consensus report from the global clinical nutrition community. Clin Nutr. 2019 Feb;38(1):1-9. doi: 10.1016/j.clnu.2018.08.002. Epub 2018 Sep 3. PMID 30181091
- [Background] Rumsfeld JS, Alexander KP, Goff DC Jr, Graham MM, Ho PM, Masoudi FA, Moser DK, Roger VL, Slaughter MS, Smolderen KG, Spertus JA, Sullivan MD, Treat-Jacobson D, Zerwic JJ; American Heart Association Council on Quality of Care and Outcomes Research, Council on Cardiovascular and Stroke Nursing, Council on Epidemiology and Prevention, Council on Peripheral Vascular Disease, and Stroke Council. Cardiovascular health: the importance of measuring patient-reported health status: a scientific statement from the American Heart Association. Circulation. 2013 Jun 4;127(22):2233-49. doi: 10.1161/CIR.0b013e3182949a2e. Epub 2013 May 6. No abstract available. PMID 23648778
- [Background] Nieminen MS, Dickstein K, Fonseca C, Serrano JM, Parissis J, Fedele F, Wikstrom G, Agostoni P, Atar S, Baholli L, Brito D, Colet JC, Edes I, Gomez Mesa JE, Gorjup V, Garza EH, Gonzalez Juanatey JR, Karanovic N, Karavidas A, Katsytadze I, Kivikko M, Matskeplishvili S, Merkely B, Morandi F, Novoa A, Oliva F, Ostadal P, Pereira-Barretto A, Pollesello P, Rudiger A, Schwinger RH, Wieser M, Yavelov I, Zymlinski R. The patient perspective: Quality of life in advanced heart failure with frequent hospitalisations. Int J Cardiol. 2015 Jul 15;191:256-64. doi: 10.1016/j.ijcard.2015.04.235. Epub 2015 May 1. PMID 25981363
- [Background] Larsson SC, Tektonidis TG, Gigante B, Akesson A, Wolk A. Healthy Lifestyle and Risk of Heart Failure: Results From 2 Prospective Cohort Studies. Circ Heart Fail. 2016 Apr;9(4):e002855. doi: 10.1161/CIRCHEARTFAILURE.115.002855. PMID 27072861
- [Background] Kontodimopoulos N, Argiriou M, Theakos N, Niakas D. The impact of disease severity on EQ-5D and SF-6D utility discrepancies in chronic heart failure. Eur J Health Econ. 2011 Aug;12(4):383-91. doi: 10.1007/s10198-010-0252-4. Epub 2010 May 15. PMID 20473544
- [Background] Bekfani T, Pellicori P, Morris D, Ebner N, Valentova M, Sandek A, Doehner W, Cleland JG, Lainscak M, Schulze PC, Anker SD, von Haehling S. Iron deficiency in patients with heart failure with preserved ejection fraction and its association with reduced exercise capacity, muscle strength and quality of life. Clin Res Cardiol. 2019 Feb;108(2):203-211. doi: 10.1007/s00392-018-1344-x. Epub 2018 Jul 26. PMID 30051186
- [Background] Berg J, Lindgren P, Mejhert M, Edner M, Dahlstrom U, Kahan T. Determinants of Utility Based on the EuroQol Five-Dimensional Questionnaire in Patients with Chronic Heart Failure and Their Change Over Time: Results from the Swedish Heart Failure Registry. Value Health. 2015 Jun;18(4):439-48. doi: 10.1016/j.jval.2015.02.003. Epub 2015 May 16. PMID 26091598
- [Background] Balestroni G, Bertolotti G. [EuroQol-5D (EQ-5D): an instrument for measuring quality of life]. Monaldi Arch Chest Dis. 2012 Sep;78(3):155-9. doi: 10.4081/monaldi.2012.121. Italian. PMID 23614330
- [Background] Malhotra R, Bakken K, D'Elia E, Lewis GD. Cardiopulmonary Exercise Testing in Heart Failure. JACC Heart Fail. 2016 Aug;4(8):607-16. doi: 10.1016/j.jchf.2016.03.022. Epub 2016 Jun 8. PMID 27289406
- [Background] Tager T, Hanholz W, Cebola R, Frohlich H, Franke J, Doesch A, Katus HA, Wians FH Jr, Frankenstein L. Minimal important difference for 6-minute walk test distances among patients with chronic heart failure. Int J Cardiol. 2014 Sep;176(1):94-8. doi: 10.1016/j.ijcard.2014.06.035. Epub 2014 Jul 1. PMID 25049008
- [Background] Ingle L, Cleland JG, Clark AL. The relation between repeated 6-minute walk test performance and outcome in patients with chronic heart failure. Ann Phys Rehabil Med. 2014 Jun;57(4):244-53. doi: 10.1016/j.rehab.2014.03.004. Epub 2014 May 2. PMID 24835160
- [Background] Deboeck G, Van Muylem A, Vachiery JL, Naeije R. Physiological response to the 6-minute walk test in chronic heart failure patients versus healthy control subjects. Eur J Prev Cardiol. 2014 Aug;21(8):997-1003. doi: 10.1177/2047487313482283. Epub 2013 Mar 19. PMID 23513011
- [Background] Elazzazi A, Chapman N, Murphy E, White R. Measurement of distance walked and physiologic responses to a 6-minute walk test on level ground and on a treadmill: a comparative study. J Geriatr Phys Ther. 2012 Jan-Mar;35(1):2-7. doi: 10.1519/JPT.0b013e31821c91b1. PMID 22189948
- [Background] Harris KM, Krantz DS, Kop WJ, Marshall J, Robinson SW, Marshall JM, Gottlieb SS. A New Clinically Applicable Measure of Functional Status in Patients With Heart Failure: The 60-Foot Walk Test. JACC Heart Fail. 2017 Jun;5(6):411-420. doi: 10.1016/j.jchf.2017.02.005. Epub 2017 May 10. PMID 28501523
- [Background] Reeves GR, Forman DE. Gait Speed: Stepping Towards Improved Assessment of Heart Failure Patients. JACC Heart Fail. 2016 Apr;4(4):299-300. doi: 10.1016/j.jchf.2016.02.002. No abstract available. PMID 27033017
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Delmonico MJ, Harris TB, Visser M, Park SW, Conroy MB, Velasquez-Mieyer P, Boudreau R, Manini TM, Nevitt M, Newman AB, Goodpaster BH; Health, Aging, and Body. Longitudinal study of muscle strength, quality, and adipose tissue infiltration. Am J Clin Nutr. 2009 Dec;90(6):1579-85. doi: 10.3945/ajcn.2009.28047. Epub 2009 Oct 28. PMID 19864405
- [Background] Springer J, Springer JI, Anker SD. Muscle wasting and sarcopenia in heart failure and beyond: update 2017. ESC Heart Fail. 2017 Nov;4(4):492-498. doi: 10.1002/ehf2.12237. PMID 29154428
- [Background] Intwala S, Balady GJ. Physical Activity in the Prevention of Heart Failure: Another Step Forward. Circulation. 2015 Nov 10;132(19):1777-9. doi: 10.1161/CIRCULATIONAHA.115.018831. Epub 2015 Oct 5. No abstract available. PMID 26438782
- [Background] Jonkman NH, Westland H, Groenwold RH, Agren S, Atienza F, Blue L, Bruggink-Andre de la Porte PW, DeWalt DA, Hebert PL, Heisler M, Jaarsma T, Kempen GI, Leventhal ME, Lok DJ, Martensson J, Muniz J, Otsu H, Peters-Klimm F, Rich MW, Riegel B, Stromberg A, Tsuyuki RT, van Veldhuisen DJ, Trappenburg JC, Schuurmans MJ, Hoes AW. Do Self-Management Interventions Work in Patients With Heart Failure? An Individual Patient Data Meta-Analysis. Circulation. 2016 Mar 22;133(12):1189-98. doi: 10.1161/CIRCULATIONAHA.115.018006. Epub 2016 Feb 12. PMID 26873943
- [Background] Bonilla-Palomas JL, Gamez-Lopez AL, Castillo-Dominguez JC, Moreno-Conde M, Lopez Ibanez MC, Alhambra Exposito R, Ramiro Ortega E, Anguita-Sanchez MP, Villar-Raez A. Nutritional Intervention in Malnourished Hospitalized Patients with Heart Failure. Arch Med Res. 2016 Oct;47(7):535-540. doi: 10.1016/j.arcmed.2016.11.005. PMID 28262195
- [Background] Henry CJ. Basal metabolic rate studies in humans: measurement and development of new equations. Public Health Nutr. 2005 Oct;8(7A):1133-52. doi: 10.1079/phn2005801. PMID 16277825
- [Background] Harris JA, Benedict FG. A Biometric Study of Human Basal Metabolism. Proc Natl Acad Sci U S A. 1918 Dec;4(12):370-3. doi: 10.1073/pnas.4.12.370. No abstract available. PMID 16576330
- [Background] Ainsworth BE, Haskell WL, Leon AS, Jacobs DR Jr, Montoye HJ, Sallis JF, Paffenbarger RS Jr. Compendium of physical activities: classification of energy costs of human physical activities. Med Sci Sports Exerc. 1993 Jan;25(1):71-80. doi: 10.1249/00005768-199301000-00011. PMID 8292105
- [Result] Rahman A, Jafry S, Jeejeebhoy K, Nagpal AD, Pisani B, Agarwala R. Malnutrition and Cachexia in Heart Failure. JPEN J Parenter Enteral Nutr. 2016 May;40(4):475-86. doi: 10.1177/0148607114566854. Epub 2015 Jan 29. PMID 25634161